CLINICAL TRIAL: NCT05718375
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled, Parallel Phase IIb Clinical Trial for the Efficacy Assessment and Safety Evaluation by Treating CU01-1001 for 24 Weeks in Type 2 Diabetic Nephropathy Patients With Albuminuria
Brief Title: Phase IIb Clinical Trial for the Efficacy and Safety by CU01-1001 for 24 Weeks in Type 2 DM Patients With Albuminuria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Curacle Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CU01-1001-DN-P2b
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CU01-1001 (low dose) (Experimental): 1 Tab/3 times/day (CU01-1001 120 mg, Breakfast and Dinner; Placebo 120 mg, Lunch)
  Interventions: Drug: CU01-1001; Drug: Placebo
- CU01-1001 (high dose) (Experimental): 1 Tab/3 times/day (CU01-1001 120 mg, Breakfast, Lunch, and Dinner)
  Interventions: Drug: CU01-1001
- Placebo (Placebo Comparator): 1 Tab/3 times/day (Placebo, Breakfast, Lunch, and Dinner)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CU01-1001 — CU01-1001
  Arms: CU01-1001 (high dose); CU01-1001 (low dose)
Drug: Placebo — Placebo
  Arms: CU01-1001 (low dose); Placebo

SUMMARY:
To evaluate the efficacy and safety of CU01-1001 administered for 24 weeks in type 2 diabetic nephropathy patients with albuminuria.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged 30 years or above
2. Patients diagnosed as type 2 diabetes prior to screening
3. Patients receiving ACE inhibitors (angiotensin-converting-enzyme inhibitor) or ARB (angiotensin II receptor blockers) for at least 8 weeks prior to screening
4. Patients who experienced albuminuria (albumin to creatinine ratio) 200~1,000 mg/g Cr) at least twice prior to 24weeks including screening results
5. Patients with blood pressure ≤ 140/90mmHg at screening
6. Patients with 25 ≤ GFR (glomerular filtration rate) ≤ 75ml/min/1.73m2 at screening
7. Patients with 6.5% < HbA1c ≤ 9% at screening

Exclusion Criteria:

1. Patients with past medical history of acute renal failure within 12weeks prior to screening; or Increase in SCr ≥ 0.3 mg/dL within 48 hours; or an increase in SCr ≥ 1.5-fold from baseline (the lowest value) within 12 weeks; or urine output <0.5mg/kg/hour for 6 hours
2. NYHA class III~IV
3. Patients with medical history related liver disease and hepatic function as follows: ALT (alanine aminotransferase) or AST (aspartate aminotransferase) >3 X institutional upper limit of normal (ULN), or Total bilirubin >3 X institutional upper limit of normal (ULN)
4. Patients with malabsorption due to organic gastrointestinal disorder or chronic gastroenterological disorders at screening (short-bowel syndrome, active Crohn's disease, and ulcerative colitis, etc.)
5. Patients with acute disease (including infectious diseases) at screening and who are thought to be unable to participate in the clinical study)
6. Within 12 weeks of the informed consent, patients who had the diagnosis and procedures of the following cardiovascular diseases: cardiac failure (NYHA class III and IV), unstable angina pectoris, myocardial infarction, transient ischemic attack, cerebro-vascular accident, history of peripheral vascular disease or coronary artery bypass surgery, and percutaneous transluminal coronary angioplasty
7. Patients with history of alcohol or drug abuse
8. Patients with any allergic reaction to the investigational product or its components
9. Patients who are planning to receive dialysis or renal transplantation within 36 weeks (9 months) in the future
10. Patients who are expected to have lower compliance with protein-limited diets and the use of the study drug
11. Women who are pregnant or breastfeeding a baby
12. Women who are able to become pregnant and do not agree to use acceptable contraception as defined by the protocol; however, women of childbearing potential who have not gone sterility procedures can participate in the study only for negative pregnancy test, and should agree to maintain effective contraception (implants of intrauterine device or intrauterine system, double barrier contraception (condom, diaphragm, sponge or cervical cap with spermicide), oral contraceptives, sterilization, and total abstinence) throughout the study
13. Patients who participated in other clinical study within 12 weeks of the participation in this study
14. Patients who are not eligible for this study participation in the judgment of the principal investigator or sub-investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change rate of urinary albumin/creatinine ratio (UACR) at 24 weeks compared to baseline | Day 0, 24 weeks
  Change rate of urinary albumin/creatinine ratio (UACR) at 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: KyuChang Won, Principal Investigator — Yeongnam University Medical Center; HyeJin Yoo, Principal Investigator — Koera University Guro Hospital; Jun Hwa Hong, Principal Investigator — Eulji University Hospital; Young Min Cho, Principal Investigator — Seoul National University Medical Center
Locations (1):
- Yeongnam University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No